CLINICAL TRIAL: NCT00423384
Title: Ibandronate Versus Placebo as add-on to Active Vitamin D and Calcium in the Prevention of Bone Loss After Renal Transplantation.
Brief Title: Ibandronate Versus Placebo in the Prevention of Bone Loss After Renal Transplantation.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Smerud Medical Research International AS (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Knut Smerud, Smerud Medical Research International AS
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMR-1471; EUDRACT no.: 2006-003884-30
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2010-03

CONDITIONS: Renal Transplant
Keywords: Ibandronate; Placebo; Doubleblind; Bone; loss; Kidney; transplant
MeSH Terms: interventions — Ibandronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Ibandronate
  Interventions: Drug: Ibandronate
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: 2
Drug: Ibandronate — I.v.
  Arms: 1

SUMMARY:
Loss of bone mass is a common complication in patients with end-stage-renal failure, both before and particularly after transplantation. In addition to standard underlying therapy with calcium and active vitamin D, we will study the effect of ibandronate (a bisphosphonate) versus placebo on bone mineral density as well as incidence of fracture rates after kidney transplantation.We also wish to study whether any prevented bone loss will also lead to reduced cardiovascular disease. Patients will be followed for 12 months after transplantation, and the ibandronate treatment is one injection every 3 months.

DETAILED DESCRIPTION:
Demographic, medical history, previous and current medication, as well as baseline measurements of Bone Mineral Density (BMD), laboratory efficacy and safety variables as well as Quality-of-Life scores will be undertaken in the period from 1 week prior to transplantation until 1 week after transplantation. In this period, any existing fractures will be determined using traditional x-ray of the thoraco-lumbar columna. Renal graft functioning as well as transplantation complications will be followed tightly, and calcium supplementation as well as active vitamin D (calcitriol) will be administered together with the standard immunosuppressive regimen.

As soon as patients have recovered from transplantation, and renal functioning is considered sufficiently stable, and no later than 28 days after the transplantation, qualified patients will be randomised to receive either ibandronate or placebo, stratified by gender. Bone mineral density and most of the clinical data and laboratory tests will then be followed until 12 months after transplantation as described in the attached flowchart (section 11.1), with hospital visits for administration of study drugs and follow-up of at 13, 26, 39 and 52 weeks after transplantation. Furthermore, all the patients will be followed prospectively from the time of transplantation and for ten years with regard to cardiovascular events. Data concerning cardiovascular events will be collected from the Norwegian renal registry for the whole study population in the follow up period of about 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipients
* Adults, ≥ 18 years of age
* Either gender
* Signed informed consent

Exclusion Criteria:

* Persisting s-Ca > 2.55 mmol/L (through the first two weeks after transplantation)
* Impaired graft functioning (estimated GFR <30 ml/min)
* Previous (within the last 12 months) treatment with bisphosphonates, sodium fluoride, calcitonin, strontium, PTH, SERM, growth hormone or anabolic steroids at any time before transplantation.
* Known adynamic bone disease
* Previous parathyroidectomy
* Pregnant or lactating females or females of childbearing potential who do not use an approved method of contraception (oral contraceptives or IUD); positive urine pregnancy test, where applicable.
* Use of any investigational drug (s) and/or device(s)
* Previous participation in this trial
* History of hypersensitivity to bisphosphonates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Difference in percent lumbar BMD change from baseline to 12 months between the two treatment groups. | December 2010

SECONDARY OUTCOMES:
Lumbar BMD change; absolute and relative | December 2010
Hip BMD change; absolute and relative | December 2010
Radial BMD change; absolute and relative | December 2010
Femural BMD change; absolute and relative | December 2010
Change in height | December 2010
Change in biochemical efficacy and bone markers | December 2010
Change in HRQoL scores (SF-36 and mini OQOL) | December 2010
Incidence of post-transplant complications | December 2010
Frequency of clinically significant safety laboratory variables | December 2010
Adverse event rates | December 2010

CONTACTS AND LOCATIONS:
Overall Officials: Knut T Smerud, MSc, Study Director — Smerud Medical Research International AS, Drammensveien 41, N-0271 Oslo, Norway
Locations (1):
- Rikshospitalet-Radiumhospitalet Medical Center, Oslo, Norway

REFERENCES:
- [Derived] Strommen RC, Godang K, Hovd MH, Finnes TE, Smerud K, Hartmann A, Asberg A, Bollerslev J, Pihlstrom HK. Hip geometry and strength remain stable the first year after kidney transplantation-an ibandronate/placebo post hoc analysis. JBMR Plus. 2024 Oct 24;8(12):ziae130. doi: 10.1093/jbmrpl/ziae130. eCollection 2024 Dec. PMID 39588131